CLINICAL TRIAL: NCT04537182
Title: Surgical Compared to Bronchoscopic Lung Volume Reduction in Patients With Severe Emphysema: an International Multi-center Randomized Controlled Trial
Brief Title: Surgical Compared to Bronchoscopic Lung Volume Reduction in Patients With Severe Emphysema
Acronym: SINCERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isabelle Opitz, Professor, MD (Other)
Responsible Party: Sponsor-Investigator, Isabelle Opitz, Professor, MD, Prof. MD, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SINCERE
Record Dates: First submitted 2020-08-20; First posted 2020-09-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Emphysema
Keywords: LVRS; BLVR; endobronchial valves; heterogeneous empyhsema; non-heterogeneous emphysema
MeSH Terms: conditions — Emphysema | interventions — Pneumonectomy

STUDY DESIGN:
Intervention Model Description: International, multi-center, open label, morphology- and site-stratified, 1:1 randomized, actively controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LVRS treatment group (Experimental): A bilateral lung volume reduction surgery (LVRS) by video-assisted thoracoscopic surgery (VATS) is performed under general anesthesia with double lumen endobronchial intubation. Unilateral treatment is accepted in cases with severe adhesions or intraoperative instability making a bilateral procedure unsafe.
  Interventions: Procedure: Lung volume reduction surgery
- BLVR study group (Active Comparator): Unilateral bronchoscopic lung volume reduction with endobronchial valves (EBV) is performed using a flexible bronchoscope under general anesthesia and under full attendance of an anesthesiologist. Valves are placed unilaterally in segmental or subsegmental bronchi in the target lobe with the goal of complete atelectasis.
  Interventions: Procedure: Bronchoscopic lung volume reduction with valves

INTERVENTIONS:
Procedure: Lung volume reduction surgery — Lung volume reduction by surgery
  Other Names: LVRS
  Arms: LVRS treatment group
Procedure: Bronchoscopic lung volume reduction with valves — Lung volume reduction with endobronchial valves.
  Other Names: BLVR
  Arms: BLVR study group

SUMMARY:
The investigators plan to perform a randomized controlled trial that compares bilateral lung volume reduction surgery (LVRS) with bronchoscopic lung volume reduction (BLVR) using endobronchial valves in terms of efficacy and patient safety.

DETAILED DESCRIPTION:
Advanced lung emphysema has a considerable impact on quality of life in patients with chronic obstructive pulmonary disease. There are positive reports of surgical as well as bronchoscopic volume reduction in selected patients, but data comparing LVRS and BLVR is unfortunately lacking to date. The investigators therefore anticipate that their study will make an important contribution to the worldwide efforts in better understanding selection and management of surgical and bronchoscopic treatment of emphysema patients and that it will be of high public interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from emphysema (all morphologies, uni- or bilateral distribution) potentially qualifying for both study procedures, LVRS or BLVR (if possible, perfusion scintigraphy within < 6 month of screening, CT scan within < 4 months of screening)
* Age ≥ 30 and ≤ 80 years
* Body Mass Index (BMI) ≥ 16, but ≤ 35 kg/m2
* Non-smoking for 3 months prior to screening interview
* Patient is able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* FEV1 more than 50% predicted
* TLC less than 100 % predicted, RV less than 175% predicted, RV/TLC less than 58% predicted, and DLCO ≤ 20% predicted in homogeneous emphysema and DLCO ≤ 15% in heterogeneous emphysema, respectively
* PaO2 ≤ 6.0 kPa (45mm Hg) at ambient air (only applicable for homogeneous morphology!)
* PaCO2 ≥ 6.6 kPa (50 mmHg) at ambient air (only applicable for homogeneous morphology!)
* Patients with incomplete interlobar fissures as revealed by quantitative computed tomography analysis with StratX® (fissure completeness ≤ 80%)
* Patients with collateral ventilation as evidenced by bronchoscopic Chartis® measurement (only performed if fissure completeness according to StratX® is < 95%)
* 6-minute walking distance ≥ 470m
* More than two COPD exacerbation episodes requiring hospitalization in the last year
* More than two instances of pneumonia episodes in the last year
* Unplanned weight loss ≥ 10% within 90 days prior to enrollment
* Pulmonary hypertension as evidenced by Delta Psyst RV-RA > 35 mmHg on recent echocardiography (within 3 months prior to screening) and confirmed by RHC (mPAP ≥ 35 mmHg) and signs of moderate to severe RV dysfunction.
* Evidence of left ventricular ejection fraction (LVEF) less than 45% on recent echocardiography (within 3 months prior to screening)
* History of exercise-related syncope
* Myocardial infarction or congestive heart failure within 6 months of screening
* Clinically significant arrhythmias that might put the patient at risk in regard to the interventions
* Prior LVR (any method), bullectomy, or lobectomy
* Clinically significant bronchiectasis with expectoration of ≥ 2 tablespoons/day.
* Pulmonary nodule requiring surgery
* Unable to safely discontinue anticoagulants or dual antiplatelet therapy for 7 days
* Patients with a life expectancy of less than one year

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline value in FEV1 (ml) | 6 months after intervention
  Percent change in FEV1

SECONDARY OUTCOMES:
Change from baseline value in FEV1 | 3 and 12 months after intervention
  Percent change in forced expiratory volume (FEV1)
Change from baseline value in RV | 3, 6 and 12 months after intervention
  Percent change in residual volume (RV)
Change from baseline value in TLC | 3, 6 and 12 months after intervention
  Percent change in total lung capacity (TLC)
Change from baseline value in RV/TLC | 3, 6 and 12 months after intervention
  Percent change in RV-to-TLC ratio
Change from baseline value in DLCO | 3, 6 and 12 months after intervention
  Percent change in diffusion capacity (DLCO)
Change from baseline value in 6-minute walking distance | 3, 6 and 12 months after intervention
  Distance that can be walked within 6 minutes
Change from baseline value in mMRC dyspnea score | 3, 6 and 12 months after intervention
  Degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4
Change from baseline in quality of life (SGRQ, EQ-5D-5L) | 3, 6 and 12 months after intervention
  St. George's Respiratory Questionnaire to assess quality of life
Change from baseline regarding pain (PDI score) | 3, 6 and 12 months after intervention
  Pain Disability Index score
Change from baseline regarding pain (VAS) | 3, 6 and 12 months after intervention
  Pain assessment with visual analog scale (VAS)
Incidence of (serious) adverse events / re-interventions | 3, 6 and 12 months after intervention
  Number and degree of adverse events after intervention
30-days mortality | 1 month
  Number of deaths (all causes) 1 month after intervention
90-days mortality | 3 months
  Number of deaths (all causes) 3 months after intervention
Overall survival rate | 12 months
  Percentage of patients alive 1 year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Opitz, Prof. MD, Principal Investigator — University of Zurich
Locations (6):
- Universitätsklinik für Thoraxchirurgie, Medical University of Vienna, Vienna, Austria
- University Hospital Leuven, Leuven, Belgium
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- Switzerland (3):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Lausanne University Hospital (CHUV), Lausanne, Canton of Vaud
  - University Hospital Zurich, Division of Thoracic Surgery, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No